CLINICAL TRIAL: NCT05449496
Title: Dietary Intervention to Improve Kidney Transplant Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1771192
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant; Complications; Kidney Diseases; Transplant;Failure,Kidney; Diabetes; Hypertension; Obesity; Diet, Healthy; Lifestyle, Healthy
Keywords: diet
MeSH Terms: conditions — Kidney Diseases; Diabetes Mellitus; Hypertension; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Dietary Education Curriculum

INTERVENTIONS:
Behavioral: Dietary Education Curriculum — Curriculum of dietary education and group-based counseling to encourage whole-food plant-based eating
  Arms: Intervention

SUMMARY:
Randomized controlled trial of a curriculum intervention teaching patients to eat a whole-food plant-based dietary pattern versus standard of care in kidney transplant recipients within the first few months of transplant

DETAILED DESCRIPTION:
A whole-food plant-based dietary pattern has emerged as fundamental in preventing and treating many of the lifestyle-related diseases of Western medicine, including cardiovascular disease, diabetes, hyperlipidemia, obesity, hypertension, chronic kidney disease and certain cancers. These diseases often occur or recur in the post-transplant population, leading to patient and graft loss. However, dietary education for kidney transplant recipients is not standardized and many patients remain ignorant about optimum healthy dietary practices. These patients are further challenged by the common occurrence of electrolyte derangements that require dietary restrictions. We propose a randomized controlled trial of a dietary intervention that focuses on whole-food plant-based eating in the kidney transplant population, testing this dietary pattern's impact on recipient health outcomes. This study addresses the critical need for cost-effective and safe strategies to improve health outcomes in transplant recipients and preserve kidney graft function. We have assembled an interdisciplinary team with expertise in transplant nephrology, lifestyle medicine, plant-based renal nutrition, health coaching and biostatistics to investigate the following aims: (1) to test the efficacy of a whole-food plant-based diet on improving kidney recipient cardiovascular and metabolic health and kidney allograft function, (2) to test the effect of a whole-food plant-based diet on kidney recipient post-transplant complication rates, and (3) to test the feasibility of a dietary education program on kidney transplant recipients' ability to adhere to a whole-food plant-based diet, all within a 12-month randomized controlled trial of plant-based diet versus usual care. Dietary counseling will focus on eating a predominantly plant-based diet comprised of fruits, vegetables, whole grains and legumes, and low in animal products, fats and processed foods. Dietary counseling will occur in group-based sessions weekly for the first month, then biweekly for 5 months. Patients will be followed for 12 months. This study has the potential to establish dietary intervention as a way to prolong kidney graft survival and to improve overall health and survival in kidney transplant recipients. This study will also launch a cohort of patients whose dietary patterns can be followed and compared over time, providing groundwork for further research into the connections between diet and kidney-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient aged 18 or greater
* Post-transplant months 2-12
* eGFR >= 20 mL/min
* Have at least one of the following:

  1. Hypertension history (BP >= 150/90 or on BP medications)
  2. Hyperglycemia history (FBG >= 100 x 2 or on diabetes medications)
  3. Overweight (BMI >= 25)

Exclusion Criteria:

* Rejection episode before study enrollment
* Gastrointestinal feeding tube or requires alternative nutrition
* Unable to understand or read English
* Unable to attend online classes or complete study questionnaires independently
* Already eating a plant-based diet
* Unwilling to make dietary changes
* Pregnant or breastfeeding
* Unable to consent
* Blindness
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiometabolic health measures | 1 year
  Proportion of individuals achieving normotension, normoglycemia and weight reduction
Post-transplant complications rates | 1 year
  Composite incidence of emergency medical visits, hospitalizations and infections

SECONDARY OUTCOMES:
Dietary complications | 1 year
  Incidence of diarrhea, use of electrolyte correcting medications, severity of hyper- and hypoglycemic events

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided